CLINICAL TRIAL: NCT05484973
Title: A Post-market Multi-center Prospective Study to Assess the Ability of the Portable Scalp Cooling System (PSCS) to Prevent Hair Loss in Women Receiving Specific Chemotherapy Regimens for Breast Cancer Stages I-III.
Brief Title: Study to Assess the Ability of the Portable Scalp Cooling System (PSCS) to Prevent Hair Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cooler Heads Care Inc. (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: COOL-CLIN-2022-01
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Alopecia; Chemotherapy-induced Alopecia; Hair Loss; Breast Cancer
MeSH Terms: conditions — Alopecia; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All patients will use AMMA (Experimental): Device: AMMA Portalbe Scalp Cooling System AMMA is indicated for use in chemotherapy infusion centers, during transit from the infusion center andat home and is intended for use by patients who are undergoing chemotherapy treatment and who want to reduce the likelihood of chemotherapy-induced alopecia.
  Interventions: Device: AMMA Portalbe Scalp Cooling System

INTERVENTIONS:
Device: AMMA Portalbe Scalp Cooling System — AMMA Portalbe Scalp Cooling System AMMA is indicated for use in chemotherapy infusion centers, during transit from the infusion center andat home and is intended for use by patients who are undergoing chemotherapy treatment and who want to reduce the likelihood of chemotherapy-induced alopecia.

SUMMARY:
The purpose of this prospective study is to assess the ability of AMMA to prevent hair loss in women receiving chemotherapy (CT) for early-stage breast cancer. Additionally, the purpose is also to assess the safety, tolerability and compliance, quality of life, and satisfaction with hair preservation after CT treatment.

DETAILED DESCRIPTION:
This is a prospectively enrolling, post-market, on-label study to assess the ability of the AMMA PSCS to prevent hair loss in women receiving CT for early-stage breast cancer, and to assess the safety, tolerability and compliance, patient quality of life, and satisfaction with hair after treatment. Female patients at least 21 years of age with stage I, II, or III breast cancer who are receiving a taxane-containing CT regimen that is scheduled to be completed within six months will be identified and data from the electronic health record (EHR) as well as prospective data will be collected.

AMMA is designed to be used by patients in the chemotherapy infusion center, during transport from the infusion center to home, and after arrival at home. Patients will participate in training in AMMA use and will be asked to bring the device to the chemotherapy infusion center for use during each chemotherapy treatment visit. The device will be used for 30 minutes prior to the start of chemotherapy, during chemotherapy and for at least 2.5 hours after chemotherapy. Scalp photos will be obtained at baseline and after the last chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients ≥ 21 years of age
2. Documented diagnosis of breast cancer, stage I, II, or III
3. A planned taxane-containing CT regimen in the adjuvant or neoadjuvant setting with curative intent
4. Concomitant agents may include trastuzumab, pertuzumab, or other CT agents such as cyclophosphamide, or carboplatin Note: Targeted and/or hormonal therapies intended for use after completion of the taxane-containing CT regimen will not be considered part of the study treatment period, and the AMMA PSCS will not be used during the post-CT targeted and/or hormonal therapy period
5. Plan to complete the current CT regimen within six months
6. At least two years out from the last CT causing hair loss with complete recovery of hair
7. Karnofsky17 performance status 80% or greater
8. Willing and able to sign informed consent for this study
9. Willing and able to complete all required study procedures

Exclusion Criteria:

1. Patients with female pattern baldness resembling picture I-3 or higher on the Savin scale
2. Autoimmune disease affecting hair; e.g. alopecia areata, systemic lupus with associated hair loss, others
3. A history of whole brain radiation
4. Plans to use a CT regimen other than those specified in the inclusion criteria; specifically, a regimen not including paclitaxel or docetaxel or a regimen including an anthracycline (AC/T, EC/T, TAC, etc.)
5. Hormone therapy concurrent with CT. Hormone therapy after CT is permitted
6. Current and/or prior use of hair growth products, such as Nutrafol, minoxidil, and Keranique
7. A serious concurrent infection or medical illness which would jeopardize the ability of the patient to complete the planned therapy and follow-up
8. History of persistent grade 2 (or higher) alopecia induced by prior chemotherapeutic regimens
9. History of and/or current exposure to other agents, drugs, device, or procedure that may cause hair loss
10. Cold sensitivity
11. Intercurrent life-threatening malignancy
12. Evidence of untreated or poorly controlled hyperthyroidism or hypothyroidism
13. History or current diagnosis of any of the following: Cold agglutinin disease, cryoglobulinemia, or cryofibrinogenemia
14. Concurrent hematologic malignancy
15. Participation in any other clinical investigation
16. Concurrent treatment with any investigational agent
17. Any reason the investigator does not believe the patient is a good candidate for the study

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 99 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Hair Loss | 3 Weeks
  To evaluate hair loss as assessed by the investigator at 3 weeks (±1 week) after the completion of the last CT treatment/infusion visit using the Common Terminology Criteria for Adverse Events (CTCAE) post-treatment, by photographs, compared to baseline photographs.

SECONDARY OUTCOMES:
Device-related adverse events | 3 Weeks
  To assess safety of the AMMA PSCS based on the occurrence of device-related adverse events, occurrence of scalp changes determined by physical examination, and patient symptoms with use of the PSCS.
Scalp changes | 3 Weeks
  Occurrence of scalp changes in patients during and after use of the AMMA PSCS.
Patient symptoms | 3 Weeks
  Patient symptoms reported during use of the AMMA PSCS as recorded by a symptom survey following each infusion session.
Subject's tolerability | 3 Weeks
  Subject's tolerability of AMMA PSCS treatment demonstrated by responses to questions related to tolerability.
Patient assessment of hair loss | 3 Weeks
  Patient assessment of hair loss as recorded in the Alopecia Self-Report Survey at post-treatment follow-up according to the following scale: <50% of normal for the patient, or ≥50% hair loss.
Patient satisfaction and QoL - Body Image Scale (BIS) | 3 Weeks
  Patient satisfaction and QoL as assessed by the BIS at baseline and posttreatment follow-up.
  The 10-item Body Image Scale was developed by Hopwood et al. in 2001 to measure affective, behavioral, and cognitive body image symptoms. Patients can indicate body image symptoms on a 4-point scale (0 "not at all" to 3 "very much"). The total score ranges from 0 to 30 and can be calculated by summing up the 10 items. A higher score means a higher level of body image disturbance
Patient satisfaction and QoL - European Organization for Research and Treatment (EORTC) QLQ-BR23 | 3 Weeks
  Patient satisfaction and QoL as assessed by the EORTC's QLQ-BR23 at baseline and post-treatment follow-up.
  All scores are linearly transformed to a 0 to 100 scale. A high or healthy level of functioning is represented by a high functional score. A high QOL is represented by a high score for global health status or QOL. More severe symptoms or problems are represented by high symptom scores or items.
Device success | 3 Weeks
  Device success is defined as ability to set up and use the AMMA device as instructed. This will be measured for each treatment and then for all treatments. If a study subject does not complete one or more of the CT visits, that does not constitute a device failure.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Dilligan, Principal Investigator — Cooler Heads Inc.
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - Carle Health, Urbana, Illinois

IPD SHARING:
Plan to Share IPD: No